CLINICAL TRIAL: NCT04490538
Title: Echocardiographic Evaluation of Right Ventricular Systolic Function by TAPSE Parameter Measured From Subcostal View Using Anatomical M-mode - Validation Clinical Study
Brief Title: Evaluation of Right Ventricular Systolic Function by TAPSE Parameter From Subcostal View
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Roman Skulec, Principal investigator, Masaryk Hospital Usti nad Labem
Other Study IDs: 284/34
Record Dates: First submitted 2020-07-19; First posted 2020-07-29 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Transthoracic Echocardiography
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Critically ill patients hospitalised at the intensive care unit indicated to echocardiographic examination.
  Interventions: Diagnostic Test: Transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Conventional transthoracic echocardiographic examination at the intensive care unit.

SUMMARY:
The purpose of this study is to validate a new echocardiographic parameter evaluating right ventricular function.

DETAILED DESCRIPTION:
The key conventional echocardiographic parameter evaluating right ventricular systolic function is the tricuspid annular plane systolic excursion (TAPSE). It is measured in apical four chamber view by conventional M-mode imaging. Other echocardiographic parameters of right ventricular systolic function (Fractional Area Change; Tricuspid Lateral Annular Systolic Velocity; Right Ventricular Index of Myocardial Performance) are evaluated in apical four chamber view as well. However, this view might not be clearly visible in the clinical setting of critical illness and subcostal view is often preferred for its higher quality. Unfortunately, conventional M-mode can not be used for measurement in this view but anatomical M-mode imaging can. Therefore, the investigators decided to evaluate whether TAPSE measured in subcostal view by anatomical M-mode (sTAPSE) correlates with conventional TAPSE and whether reliably reflects systolic right ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* All patients hospitalised in intensive care unit indicated for transthoracic echocardiography examination

Exclusion Criteria:

* Age <18 years
* Insufficient imaging quality of transthoracic echocardiography
* Refusal of echocardiographic examination by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult intensive care unit patients.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Validity of sTAPSE in prediction of right ventricular systolic dysfunction | During the intervention
  sTAPSE is a new potential echocardiographic parameter of right ventricular systolic function measurable from subcostal view.

SECONDARY OUTCOMES:
Correlation of sTAPSE with conventional TAPSE | During the intervention
  sTAPSE is a new potential echocardiographic parameter of right ventricular systolic function measurable from subcostal view.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Masaryk Hospital Usti nad Labem
Locations (1):
- Masaryk Hospital Usti nad Labem, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077